CLINICAL TRIAL: NCT01961479
Title: Development and Evaluation of an Internet-based Cognitive Behaviour Therapy for Women With Premenstrual Syndrome (PMS)
Brief Title: Treatment of Premenstrual Syndrome - Internet-based Self-help
Acronym: praemensis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Cornelia Weise, Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: praemensis_2013
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Premenstrual Syndrome (PMS)
Keywords: Premenstrual syndrome (PMS); Premenstrual Dysphoric Disorder (PMDD); Internet-based Therapy; Cognitive Behavioural Therapy (CBT)
MeSH Terms: conditions — Premenstrual Syndrome; Premenstrual Dysphoric Disorder | interventions — Spectrometry, Fluorescence; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based CBT for patients with PMS (Experimental): The therapeutical intervention follows a treatment manual consisting of 14 modules. Patients work on up to two modules every week for eight weeks in a row. Modules comprise a) psychoeducation (e.g., information about PMS and its treatment); b) cognitive strategies (e.g., identifying and modifying dysfunctional cognitions, or coping with negative affects); and c) suggestions for lifestyle changes (e.g., sports, stress reduction, or balanced diet). Aim of the iCBT is to improve coping and thus to reduce the impairment due to premenstrual symptoms.
  Interventions: Behavioral: Internet-based CBT for patients with PMS
- waiting list (Other): During the waiting period, patients receive no treatment. After a waiting time of 2 months, patients of the waitlist receive the same iCBT treatment as the experimental group.
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Internet-based CBT for patients with PMS — Internet-based cognitive-behavioural self-help treatment
  Arms: Internet-based CBT for patients with PMS
Other: Waiting list — During the waiting period, participants receive no treatment.
  Arms: waiting list

SUMMARY:
The purpose of this study is to determine whether an internet-based CBT (iCBT) is effective in reducing the impairment caused by premenstrual symptoms.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) affects millions of women during their reproductive years. The disorder presents with emotional, cognitive, behavioural, and somatic symptoms during the final premenstrual phase and subsiding a few days after menses begins. About 75% of women of reproductive age experience a mild form of PMS (Campbell, Peterkin, O'Grady, & Sanson-Fisher, 1997). The more severe form of PMS, premenstrual dysphoric disorder (PMDD; American Psychiatric Association (APA), 1994) is considered to affect up to 8% of women of reproductive age. This severe form is associated with severe disruptions in normal functioning in work, family, or social relationships (Halbreich, Borenstein, Pearlstein, & Kahn, 2003). The defining characteristics of both-PMS and PMDD- are the cyclic pattern of symptoms, which must be confirmed by prospective daily self ratings of symptoms (PMS-Diary) over two consecutive menstrual cycles (American College of Obstetricians and Gynecologists (ACOG), 2000). PMS and PMDD differ according to the number, severity, duration, and quality of symptoms.

As a first-line intervention, the ACOG suggests pharmacotherapy, in particular selective serotonin reuptake inhibitors (SSRIs; ACOG, 2000). However, the side effects of SSRIs are intolerable to many women, leading to high rates of withdrawal from treatment (Busse et al., 2009; Dimmock, Wyatt, Jones, & O'Brien, 2000). Thus, cognitive behavioural treatments (CBT) have been suggested as an additional treatment approach (Busse et al., 2009). First studies showed promising results for CBT interventions for PMS (Busse et al., 2009; Hunter et al., 2002). However, too few randomized controlled trials have carefully investigated the efficacy of CBT for PMS.

The aim of the current study is thus to develop a CBT-oriented self-help treatment programme for women suffering from PMS or PMDD. The treatment programme consists of psychoeducation (e.g., information about PMS/PMDD and its aetiology), cognitive strategies (e.g., assessing and restructuring dysfunctional cognitions), and suggestions for lifestyle changes (e.g., sports, balanced diet, relaxation). The programme is internet-delivered (iCBT) and participants work on different chapters for eight weeks in a row. In addition to written information, participants receive e-mail feedback from a psychologist on a weekly basis. Participants are required to have sufficient knowledge of German in order to be able to read the treatment materials. After a careful diagnostic assessment (including two months symptom diary), eligible patients are randomly assigned either to the treatment group or a waitlist control group. Participants assigned to the waitlist receive the treatment after the end of the waiting period (eight weeks). Follow-up assessments take place six months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling of particular diagnostic criteria: positive retrospective symptom screening & confirmation of the diagnosis by a prospective PMS-Diary over 2 menstrual cycles
* Age 18-45 years
* Internet access
* Fluency in German

Exclusion Criteria:

* Birth of a child or lactation going back to less than 3 months
* Pregnancy
* Symptoms exist less than three cycles
* Gynaecological diseases: Hysterectomy, Gynaecological cancer, Polycystic ovary syndrome, Endometriosis, Infertility
* Current diagnosis of psychosis or bipolar disorder
* Current diagnosis of eating-disorder
* Current diagnosis of average or severe depression
* Current diagnosis of somatisation disorder
* Acute suicidal tendency
* participation in psychotherapy due to premenstrual syndrome, currently or in the past
* Begin to take antidepressants or a change of the active pharmaceutical ingredient during the last three months
* Begin to take a combined oral contraceptive pill or a change of the preparation during the last three months
* Begin to take hormones or a change of the hormone supplement during the last three months
* The taking of Benzodiazepines/Antipsychotics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2013-07; Primary Completion 2017-07 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Retrospective Screening (Ditzen et al., 2011) | pre-treatment
  assessment of premenstrual symptoms based on the Diagnostic and Statistical Manual of Mental Disorders Text Revision (DSM-IV-TR) (self-rating)
Prospective PMS-Diary (Kleinstäuber et al., unpublished) | 6 months; pre-treatment to post-treatment (4 months after admission)
  prospective daily self ratings of premenstrual symptoms based on the DSM-IV-TR (self-rating)
Impairment by the premenstrual syndrome (self-developed questionnaire) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of cognitive, emotional and functional impairment by the premenstrual syndrome (self-rating)

SECONDARY OUTCOMES:
Coping with the premenstrual symptoms (self-developed questionnaire) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of coping strategies (self-rating)
Pain Coping Questionnaire (FESV; Geissner, 2003) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of PMS related coping strategies (self-rating)
Short Form Social Support Questionnaire (Fragebogen zur sozialen Unterstützung Kurzform (F-SozU K-22); Fydrich, Sommer, & Brähler, 2007) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of the availability of social support (self-rating)
Questionnaire of the assessment of the partnership quality (FPQ; Siffert & Bodenmann, 2010) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of partnership quality (self-rating)
Effort-Reward Imbalance Questionnaire (ERI-Short-form; Siegrist, Wege, Pühlhofer, & Wahrendorf, 2009) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of work strain (self-rating)
Perceived stress scale (PSS, Cohen, 1994) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of stress perception (self-rating)
The Big Five inventory (BFI-Short-form, John, Naumann, & Soto, 2008) | pre-treatment
  assessment of personality
Pain Disability Index (PDI; Dillmann, Nilges, Saile, & Gerbershagen, 1994) | 10 months; pre-treatment (during luteal phase) to post-treatment (during luteal phase, 4 months after admission) to follow-up (during luteal phase, 10 months after admission)
  assessment of the degree of daily impairment by chronic pain (self-rating)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Weise, Ph.D., Study Chair — Philipps University Marburg; Maria Kleinstäuber, Ph.D., Study Chair — Philipps University Marburg; Carolyn Janda, Ph.D.Student, Study Chair — Philipps University Marburg; Johanna N. Kues, Ph.D.Student, Study Chair — Philipps University Marburg; Gudrun Kaiser, Ph.D Student, Study Chair — Philipps University Marburg
Locations (1):
- Philipps University Marburg, Dept. of Psychology, Division of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany

REFERENCES:
- [Background] Busse JW, Montori VM, Krasnik C, Patelis-Siotis I, Guyatt GH. Psychological intervention for premenstrual syndrome: a meta-analysis of randomized controlled trials. Psychother Psychosom. 2009;78(1):6-15. doi: 10.1159/000162296. Epub 2008 Oct 14. PMID 18852497
- [Background] Campbell EM, Peterkin D, O'Grady K, Sanson-Fisher R. Premenstrual symptoms in general practice patients. Prevalence and treatment. J Reprod Med. 1997 Oct;42(10):637-46. PMID 9350019
- [Background] Dimmock PW, Wyatt KM, Jones PW, O'Brien PM. Efficacy of selective serotonin-reuptake inhibitors in premenstrual syndrome: a systematic review. Lancet. 2000 Sep 30;356(9236):1131-6. doi: 10.1016/s0140-6736(00)02754-9. PMID 11030291
- [Background] Halbreich U, Borenstein J, Pearlstein T, Kahn LS. The prevalence, impairment, impact, and burden of premenstrual dysphoric disorder (PMS/PMDD). Psychoneuroendocrinology. 2003 Aug;28 Suppl 3:1-23. doi: 10.1016/s0306-4530(03)00098-2. PMID 12892987
- [Background] Hunter MS, Ussher JM, Cariss M, Browne S, Jelley R, Katz M. Medical (fluoxetine) and psychological (cognitive-behavioural therapy) treatment for premenstrual dysphoric disorder: a study of treatment processes. J Psychosom Res. 2002 Sep;53(3):811-7. doi: 10.1016/s0022-3999(02)00338-0. PMID 12217456
- [Background] Siegrist J, Wege N, Puhlhofer F, Wahrendorf M. A short generic measure of work stress in the era of globalization: effort-reward imbalance. Int Arch Occup Environ Health. 2009 Aug;82(8):1005-13. doi: 10.1007/s00420-008-0384-3. Epub 2008 Nov 19. PMID 19018554
- [Background] Dillmann U, Nilges P, Saile H, Gerbershagen HU. [Assessing disability in chronic pain patients.]. Schmerz. 1994 Jun;8(2):100-10. doi: 10.1007/BF02530415. German. PMID 18415443
- [Background] Kleinstauber M, Witthoft M, Hiller W. Cognitive-behavioral and pharmacological interventions for premenstrual syndrome or premenstrual dysphoric disorder: a meta-analysis. J Clin Psychol Med Settings. 2012 Sep;19(3):308-19. doi: 10.1007/s10880-012-9299-y. PMID 22426857
- [Background] American College of Obstetricians and Gynecologists (ACOG). Premenstrual syndrome. Washington, DC: National Guideline Clearinghouse, 2000.
- [Background] American Psychiatric Association (APA). Diagnostic and statistical manual for mental disorders (DSM-IV). Washington, DC: American Psychiatric Press, 1994.
- [Background] Cohen S. Perceived stress scale, 1994. Retrieved August 09, 2012, from http://updates.wcupa.edu/_academics/healthsciences/stressreductioncenter/documents/perceived_stress_scale.pdf
- [Background] Ditzen B, Nussbeck F, Drobnjak S, Spörri C, Wüest D, Ehlert U. Validierung eines deutschsprachigen DSM-IV-TR basierten Fragebogens zum prämenstruellen Syndrom. Zeitschrift für Klinische Psychologie und Psychotherapie 40(3): 149-159, 2011.
- [Background] Fydrich T, Sommer G, & Brähler E. Fragebogen zur sozialen Unterstützung (F-SozU ). Göttingen: Hogrefe, 2007.
- [Background] Geissner E. Pain Coping Questionnaire FESV. Göttingen, Germany: Hogrefe, 2003.
- [Background] Siffert A, Bodenmann G. Entwicklung eines neuen multidimensionalen Fragebogens zur Erfassung der Partnerschaftsqualität (FPQ). Zeitschrift für Familienforschung, 2010.
- [Derived] Kues JN, Janda C, Kleinstauber M, Weise C. Internet-based cognitive behavioural self-help for premenstrual syndrome: study protocol for a randomised controlled trial. Trials. 2014 Dec 2;15:472. doi: 10.1186/1745-6215-15-472. PMID 25467540
- See also: Click here for more information about this study: Treatment of the Premenstrual Syndrome - Internet-based self-help — http://www.uni-marburg.de/fb04/ag-klin/forschung/pmsd/index_html
- Available data/document: Study Protocol — http://trialsjournal.biomedcentral.com/articles/10.1186/1745-6215-15-472 — Kues, J. N., Janda, C., Kleinstaeuber, M., & Weise, C. (2014). Internet-based cognitive behavioural self-help for premenstrual syndrome: study protocol for a randomised controlled trial. Trials, 15(1), 472. doi:10.1186/1745-6215-15-472